CLINICAL TRIAL: NCT00891917
Title: Evaluation of Coenzyme q10 (Liq-nol®) Efficacy in Pediatric Patients With Down Syndrome
Brief Title: Liq-NOL Efficacy in Pediatric Patients With Down Syndrome
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: no funding
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2008-0489
Record Dates: First submitted 2009-04-29; First posted 2009-05-01 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2014-01

CONDITIONS: Down Syndrome
Keywords: Down syndrome; coenzyme Q10; language function; behavior
MeSH Terms: conditions — Down Syndrome; Language; Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Syrup (Placebo Comparator): identical placebo formulation to be administered twice a day.
  Interventions: Dietary Supplement: syrup (placebo)
- Ubiquinol-10 Syrup (Active Comparator): CoQ (LiQ-NOL®) 10.0 mg/kg/d to be administered twice a day
  Interventions: Dietary Supplement: Ubiquinol-10 Syrup

INTERVENTIONS:
Dietary Supplement: Ubiquinol-10 Syrup — 10 mg/kg/day in 2 divided doses for 3 months or Placebo Syrup for 3 months
  Other Names: LiQ-NOL
  Arms: Ubiquinol-10 Syrup
Dietary Supplement: syrup (placebo) — syrup looks exactly like the Ubiquinol-10 Syrup but has no active ingredients or supplementation
  Arms: Syrup

SUMMARY:
The purpose of this study is to measure the effects of LiQ-NOL supplementation on language production using the Clinical Evaluation of Language Fundamentals test, language sampling using the mean length of utterance test, and speech articulation using the Goldman-Fristoe Test of Articulation.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled clinical study of CoQ efficacy in a crossover design. Patients will be screened, enrolled, and studied in the outpatient clinic of the Thomas Center for Down Syndrome at CCHMC. All patients will be randomly assigned to either a liquid product (LiQ-NOL®) and an identical placebo liquid. Study drug and placebo will be administered twice a day (morning and evening).

ELIGIBILITY:
Inclusion Criteria:

* Patients ranging from 6.0 years to 16 years of age.
* Patients will have proven Trisomy 21.
* Females, incapable of bearing children or capable of practicing adequate birth control methods. Abstinence will be acceptable.
* Written informed consent will be obtained from parents of all subjects prior to enrollment. Verbal assent will be obtained from all patients with DS who have sufficient decision making ability and are at least 11 years old.

Exclusion Criteria:

* Patients who have insufficient mental and/or motor capacity to complete testing measures.
* Patients less than 6 years or older than 16 years of age.
* Patients receiving CoQ supplementation within one month prior to the study.
* Patients with evidence of disease which may adversely affect CoQ absorption, e.g. chronic diarrhea or inflammatory bowel disease.
* Patients participating in other research studies or having exposure to investigational drugs within one month prior to this study.
* Females, capable of bearing children, who are unsure of their pregnancy status or not practicing adequate birth control methods.
* Females who are pregnant.
* Patients with a known allergy to CoQ.
* Patients receiving drug treatment which is know to affect CoQ, e.g. cholesterol-lowering drugs such as "statins".

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2005-01; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To measure the effects of LiQ-NOL on language skills, expressive language ability, and speech articulation. | beginning and end of 3 month treatment period

SECONDARY OUTCOMES:
To evaluate the effects of LiQ-NOL on child behavior. | beginning and end of 3 month treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Michael V Miles, Pharm.D., Principal Investigator — Childrens Hospital Medical Center, Cincinnati; Francis Hickey, M.D., Principal Investigator — Childrens Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Miles MV, Patterson BJ, Chalfonte-Evans ML, Horn PS, Hickey FJ, Schapiro MB, Steele PE, Tang PH, Hotze SL. Coenzyme Q10 (ubiquinol-10) supplementation improves oxidative imbalance in children with trisomy 21. Pediatr Neurol. 2007 Dec;37(6):398-403. doi: 10.1016/j.pediatrneurol.2007.08.003. PMID 18021919
- [Background] Miles MV, Patterson BJ, Schapiro MB, Hickey FJ, Chalfonte-Evans M, Horn PS, Hotze SL. Coenzyme Q10 absorption and tolerance in children with Down syndrome: a dose-ranging trial. Pediatr Neurol. 2006 Jul;35(1):30-7. doi: 10.1016/j.pediatrneurol.2005.11.004. PMID 16814082